CLINICAL TRIAL: NCT07160764
Title: Evaluation of Performance and Safety of Hyalosem Cross-linked Hyaluronic Acid Adhesion Barrier Gel in Preventing Intra-uterine Adhesion Formation After Operative Hysteroscopy: A Retrospective Study
Brief Title: Safety and Performance of the Semical Adhesion Barrier Gel for Prevention of Intra-uterine Adhesion
Acronym: SEMFERTIL
Status: Not yet recruiting | Type: Observational
Sponsor: Semikal Technology (Industry)
Collaborators: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SEMFERTIL
Record Dates: First submitted 2025-08-15; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Intrauterine Abnormalities in Infertility; Asherman Syndrome; Intra-uterine Adhesions; Postoperative Adhesion of Uterus; Asherman's Syndrome
Keywords: intrauterine abnormalities; asherman's syndrome; intrauterine adhesions; postoperative adhesions
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-linked hyaluronic acid based adhesion barrier gel: Operative hysteroscopy plus adhesion barrier gel
- Control group (none): Operative hysteroscopy alone as control group

SUMMARY:
The aim of this study was to obtain short- and long-term performance and safety data of cross-linked hyaluronic acid-based adhesion barrier gel used to prevent intrauterine adhesion formation.

DETAILED DESCRIPTION:
This study was designed as a non-interventional (observational), comparative, retrospective and single-center study. The investigational device has the CE mark under 93/42/ EEC Medical Device Directive and is used in accordance with the intended use declared by the manufacturer in the user manual. Therefore, the study is a post-marketing clinical follow-up (PMCF) study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 and over
* Patients who were treated with operative hysteroscopy for intrauterine pathology (endometrial polips, myomas with uterine cavity deformation, uterine septa, intrauterine adhesion, ovarian cyst, endometrial cyst, etc.)
* Patients who had undergone operative hysteroscopy at least 30 days and at most 6 months ago
* Patients who had second-look office hysteroscopy at least once after an operative hysteroscopy

Exclusion Criteria:

* Children and adolescents under 18 years of age
* Having a body weight of more than 100 kg
* Surgeries complicated by excessive bleeding; estimated blood loss of more than 100 cc
* Surgeries complicated with uterine perforation
* Presence of uncontrolled diabetes, coagulation disorders, and other severe chronic disorders
* Presence of malignant tumor or diagnosis of cancer, presence of uterovaginal prolapse
* Concomitant peritoneal grafting or tubal implantation
* Concomitant intrauterine device implantation
* Patients without second-look hysteroscopy

According to the GDPR and clinical investigation legislation, written informed consent is not mandatory in retrospective studies as long as the patient's personal information is censored.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — biological females
Study Population: Female patients ages 18 years and over who are at risk of postoperative adhesion formation after operative hysteroscopy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of post-operative intrauterine adhesions at second look hysteroscopy | 6 months
  Incidence and severity (according to AFS classification) of intrauterine adhesions after operative hysteroscopy identified at follow-up diagnostic hysteroscopy

SECONDARY OUTCOMES:
Improvement in menstrual pattern | 6 months
  from baseline to second look hysteroscopy
Adverse events | through study completion
  Incidence and severity of the adverse events associated with adhesion barrier use

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Training and Research Hospital Gynecology and Obstetrics Clinic, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not allowed by locak regulations